CLINICAL TRIAL: NCT02527499
Title: The Effects of Combining Modified ride-on Cars With Bimanual Training on Enhancing Mobility, Socialization, Motor Function and Participation in Toddlers With Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMRPD3E0311
Record Dates: First submitted 2015-07-08; First posted 2015-08-19 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2017-01

CONDITIONS: Children With Mobility Disabilities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ROCBT group (Experimental): The participant's performance is indicative of the extent to which early power mobility training is feasible for 1 to 3 years old and diagnosed as motor delay (>1.5 sd). Parents/caregivers and occupational therapists will be responsible for Ride-On Cars with Bimanual Training Program (ROCBT) group.
  Interventions: Behavioral: Ride-On Cars with Bimanual Training Program (ROCBT)
- Early Mobility Training group (Active Comparator): The participant's performance is indicative of the extent to which early power mobility training is feasible for 1 to 3 years old and diagnosed as motor delay (>1.5 sd). Parents/caregivers and occupational therapists will be responsible for Early Mobility Training Program group.
  Interventions: Behavioral: Early Mobility Training Program
- Regular Therapy group (Active Comparator): The participant's performance is indicative of the extent to which early power mobility training is feasible for 1 to 3 years old and diagnosed as motor delay (>1.5 sd). Parents/caregivers and occupational therapists will be responsible for Regular Therapy Program group.
  Interventions: Behavioral: Regular Therapy Program

INTERVENTIONS:
Behavioral: Ride-On Cars with Bimanual Training Program (ROCBT) — The car driving training includes 2 phases: I-car exploration and II-prompted driving. Participants can learn how to move and stop the car in the car exploration phase. Through prompted driving in phase II, they can use the car as a mean to explore environments (e.g., to the elevator, to different stores) and contact with people (e.g., drive to the caregiver and get the toy). Bimanual training involves activities which include perceptual motor tasks (e.g., smear both hands with color), holding and manipulative tasks (e.g., cutting toy vegetables or fruits), posture and balance (e.g., pull a cart), and self-care and activities of daily living (e.g., drinking water from a cup with two handles).
  Arms: ROCBT group
Behavioral: Early Mobility Training Program — Most of the guidelines are similar with ROCBT, except for the bimanual training. The therapist and family will merely focus on independent mobility training and improving socialization. The training time and period is the same as ROCBT.
  Arms: Early Mobility Training group
Behavioral: Regular Therapy Program — The regular therapy group will continue the regular therapy, including physical, occupational and speech therapy. The general propose of the training is to improve the developmental scales, mobility, socialization and upper limb use in functional tasks. The research team will videotape the child's natural play and driving performance at the hospital for 1 hour/per session, 1 session/per week during the 9-week intervention phase.
  Arms: Regular Therapy group

SUMMARY:
The four purposes of this study are: 1) to examine the feasibility of combining modified ride-on cars with bimanual training (ROCBT) on mobility, socialization and motor function in toddlers with disabilities; 2) to quantify whether toddlers with disabilities are able to have more manual explorations and social interactions with ROCBT through observation and wrist-worn accelerometers; 3) to determine the critical factors of using the modified ride-on toy car on family perceptions and participation.

Independent mobility is believed to be essential for perceptual-motor, cognition, language and social skill development. It is important to increase independent mobility in toddlers with disabilities and further enhance their development, especially socialization. Assistive and power mobility devices allow toddlers with disabilities to move independently within their environment and may increase the opportunities to explore and interact with people and environment. However, issues to consider before prescribing an assistive device include factors such as age, accessibly to community environments, cost, and social acceptance of the device and the adaptability of the device to growth. To address these limitations and meet toddlers' needs, the concept of using modified ride-on toy cars in therapy becomes a novel application. Study has demonstrated the use of toy cars enhanced a child's motivation, socialization and family participation. This study is further to combine the use of customized, modified ride-on toy cars with bimanual training, to enhance the independent mobility, manual exploration and socialization through low-cost, family-centered approach. It will also improve family's understanding of children's capabilities, which improve their development.

Investigators will recruit 75 children with who are between 1 to 3 years old and diagnosed as motor delay (>1.5 sd). They will be randomly assigned to one of the following three groups: ROCBT treatment group, early mobility training group and regular therapy group. The whole study duration will be 18 weeks, including 9-week intervention and 9-week follow-up; the total amount of treatment will be equal for two groups. Standardized assessments are provided for a total of three times during the study, including the time before and after the intervention and in the end of the follow-up phase. The ROCBT and early mobility training programs will be administered by the therapist and include 120 minutes/per session, 2 sessions/per week. The research team will visit the hospital once/per week to provide 60 minutes videotaping and wearing wrist-worn accelerometers. The regular therapy group will continue their regular therapy without any additional car driving training. The research team will visit them once/per week for the assessments. The assessments include standardized measurements and behavior coding from the videotapes and accelerometers. The findings of this study will help to understand the feasibility and effectiveness of combining the low-tech modified ride-on cars with bimanual training on advancing children's mobility and socialization. They can be used in the clinic or school and are a low cost alternative or addition to other mobility devices. They may provide a novel therapeutic tool to improve mobility, socialization, family participation and development.

DETAILED DESCRIPTION:
Spontaneous self-initiated actions have consequences, and experiencing these is very educational. Independent mobility is believed to be essential for perceptual-motor and social skill development. Self-produced locomotion is an organizer of psychological changes in children with typical development, especially developmental changes in perceptions, social understanding, spatial cognitive, and emotions. In addition, through active manual exploration, children can detect the object and individual's information that relates size, orientation, shape, substance to their perceptual and movement capabilities and interpersonal relationships. Children require exploratory behaviors to gather relevant information for a task. They can learn the relationship between the object-surface and movements through increased independent mobility and manual exploration. There is convincing evidence that the use of powered mobility for children with disabilities has positive impacts on their overall development and increases their exploration. Studies are focusing on reducing the limitations in the areas of social, cognitive, perceptual, and functional development that were induced by lack of independent mobility in early ages. Limited evidence also demonstrated that early powered mobility training had positive impacts on the family participation, including decreasing parents' level of stress and increasing their satisfaction with their child's sleep patterns, ability to move out, and ability to interact and socialize with the family.

Pediatric rehabilitation, through training and assertive technology (AT), seeks to provide children with disabilities with the same level of mobility, exploration, socialization and participation for children with typical development (TD). Proponents of powered vehicles for very young children present strong reasons for introducing powered mobility to children at a time in their developmental pattern that coincides as closely as possible to when they would have begun independent mobility as a child with TD. Research has suggested that there is no negative influence on motor development or self-care abilities. In addition, children with disabilities may be more motivated to participate in therapy and may demonstrate increased head, trunk and arm-hand control for exploration in the surrounding environment. However, up to date, the lack of rigorous studies and limited evidence of the increased independent mobility and early child development across all three International Classification of Functioning, Disability and Health (ICF) levels, still signify the needs of considering early power mobility as a feasible intervention in the clinical settings for very young children who have not yet achieved a means of independent mobility and are unlikely to achieve it.

There are many basic barriers to achieving this high standard and no single AT or combination of AT can currently provide the level of mobility and exploration that children, families and therapists desire. Currently, the most critical barrier to including power mobility in EI programs is the lack of readily available power chairs for children younger than 2-3 years of age, the period when mobility is rapidly developing for children with typical development. Certain characteristics of the most common commercial pediatric power wheelchairs limit their use in the home and community spaces such as playgrounds. These limitations include price (e.g., typically >$5000), size and weight (e.g., typically >150 lbs), transportation requirements (e.g., van or truck), maintenance and aesthetics and social acceptance. Experimental power mobility devices (PMD) have the potential to address some of these limitations such as size, weight and infant use. Unfortunately these are likely years from commercial availability. Moreover, power wheelchairs have historically been designed to address a limited set of goals related to mobility with minimal consideration of socialization. Investigators believe there is a need for readily available mobility options for immediate use by very young children and their families that address some of the above limitations while expanding the role of PMD past simply mobility and into socialization.

There are four strengths of using ride-on toy cars for mobility. First, the cost is comparable or less than most mobility devices. Second, most are relatively lightweight, small and easily transported in contrast to power chairs. Third, the child-friendly, colorful toy designs are more acceptable to adults and children and likely seen as simply a toy. This may be an important aspect for clinicians wanting to start early power mobility training with families hesitant to discuss powered chair options. Fourth, because toy cars are simple electromagnetically devices, they can be modified quickly and easily to match the child's current and/or future abilities and goals. The use of modified ride-on toy cars may provide a readily available, convenient and fun way for families, therapists and early educators to help young children improve their mobility starting within the first years of life.

From our initial pilot results, it indicated that this early powered mobility training through the use of modified toy cars might enhance cognition, language, mobility, and socialization in toddlers with mobility impairments. However, the fine and gross motor remained at a similar level before and after 9-week intervention. These initial findings suggest a number of important points: 1) early power mobility training may increase exploratory behaviors and benefit independent mobility, cognitive and social development; 2) the improvements of children's development and caregiver's involvement in the training may decrease family stress level and increase family participation; 3) simple early power mobility training may not be enough to improve motor function. Better postural control coupled with reaching and grasping ability allows infants to independently explore objects in new ways for sustained periods through mouthing and touching. The seat adjustments (e.g., a seat belt er, a hip strap) of ride-on toy cars may provide sufficient postural stability for the child with disabilities, however, the impaired reaching and grasping ability may decrease the opportunities of doing manual exploration for both hands. Most daily activities are functional tasks and may require two hands doing different actions. The development of increased functional independence requires use of both hands in cooperation. Gordon et al. had asked caregivers to identify goals for the intervention, and measured the progress using goal-attainment scale (GAS). Nearly 85% of the goals were bimanual. Principles of motor learning (practice specificity) suggest the most functional way to balance the cortical activity and improve bi-manual control would be to practice bi-manual activities directly.

Bi-manual training is an approach often used by clinicians treating the upper extremity function. It appears to be better for improving bi-manual coordination and goal performance. Andersen et al. suggested that bi-manual training may be better for a child with mild impairments, or for a child without grasping abilities in one hand as tasks can be graded such that the hand can be used as passive assist to begin. Most importantly, bi-manual activities may be more motivating as they are generally more ecologically relevant and may be selected to maximize interest. Studies showed that intensive bi-manual training can significantly improve the quality and quantity of bi-manual hand use in children with hemispheric cerebral palsy (CP). It focuses on improving the coordination of both upper extremities through functional and play activities, and requires active problem solving for children to discover their bi-manual capabilities. Active discovery-learning and problem solving are principles of learning within a perception-action framework and can promote neural plasticity. Bi-manual training may allow direct practice of functional meaningful goals, and such practice can transfer to unpracticed goals and improve manual, exploratory learning.

Theoretically, using powered mobility combined with increased manual exploration as part of a comprehensive Early Intervention (EI) program within the first three years of life should not only provide mobility but also reduce secondary impairments for children with disabilities. Although of increasing interest, there is very little empirical evidence of the effects or even feasibility of early power mobility training on the family participation and overall development, particularly for mobility and socialization. Furthermore, up to date, there is no evidence on examining the effects of applying early PMD combining with bi-manual training on the active discovery-learning and upper extremity function for young children with disabilities. Our case report was the first study showing positive effects of using a ride-on car on mobility and socialization in a child with severe CP. The pilot results of the previous study also demonstrated positive impacts of implementing early ride-on car training on cognition, language, and mobility for toddlers with disabilities. It also helped to decrease the caregiver's stress level. However, motor function tended to be at the similar level before and after the 9-week intervention. In addition, little is known about the learning curve of using the PMD to improve development, e.g., at what point in time (maximal) effects are reached. Up to now, most of the studies have focused on the end results of increased amount of independent mobility in daily life. It is still unknown whether optimal (maximal) effects are being reached at all and which factors might influence the learning curve as well as the retention of treatment effects in the long term. To improve the overall development, investigators hypothesize that combining modified ride-on toy cars with bi-manual training (ROCBT) may benefit the toddler's development on cognition, socialization and motor, especially for the manual exploration. Furthermore, this combined training may improve the toddler's goal performance, enhance the family's perception on the child's capabilities and increase the function at participation level.

In this study, investigators will modify ride-on toy cars for children with disabilities for use in clinical settings as part of a 18-week power mobility training program. In addition, investigators will combine this ride-on toy use with bi-manual training and compare the results to the regular therapy. Investigators will focus on four research questions. Specifically, can investigators: 1) use the modified toy cars and combine it with bi-manual training as an effective power mobility training program to improve the exploratory behaviors and overall development; 2) select a set of dependent measures that quantify whether the children increase their exploratory behaviors; 3) determine the factors that influence family's perception on the environment, child and themselves; 4) conduct a hospital-based, power mobility training program that results in a high level of fun for the child and compliance by the family and therapists. If our results are generally positive and show significant differences among ROCBT, early powered mobility training and regular therapy, it will provide us some alternative ways either to improve the overall development or merely independent mobility and socialization. Subsequently, the future randomized controlled trial studies could further quantify the effectiveness and the feasibility with different treatment intensity and various pediatric populations.

The specific aims of this study are: 1) to examine the feasibility of combining modified ROCBT on mobility, socialization and motor function in toddlers with disabilities; 2) to quantify whether toddlers with disabilities are able to have more manual explorations and social interactions with ROCBT through observation and wrist-worn accelerators; 3) to determine the critical factors of using the modified ride-on toy car on family perceptions and participation. Through the comparison among ROCBT, early powered mobility training and regular therapy groups, investigators hypothesize that ROCBT group will have more improvements on mobility, socialization and motor functions than the early powered mobility training and the control groups. Children in the ROCBT group will have more physical activity for manual explorations and social interactions, in comparison to the early powered mobility group, due to the combined bi-manual training. In addition, investigators hypothesize that ROCBT will elicit different family perceptions on the child's capabilities and themselves, in comparison to the early powered mobility training and regular therapy.

Study Design: A pretest-post-test control group design will be applied. Three groups will be involved in this project: hospital-based, modified ride-on cars combined with bi-manual training program (ROCBT), early powered mobility training program and regular therapy program. The participants will be randomly assigned to one of the three groups by using the well-sealed, opaque envelopes when they are recruited in the study. Once the participants are recruited in the study, the research team will modify a toy car based on each participant's capabilities during this pre-intervention phase (the first two or three weeks before intervention starts), e.g., seat and steering wheel modifications. The study duration for each participant is 18 weeks, including 9-week intervention and 9-week follow-up.

Participants in the study will be 75 toddlers ages 12 months to 36 months with motor delays (sd > 1.5). They will be randomly assigned to either the powered mobility combined with bi-manual training group (25 toddlers), 25 early powered mobility training group (25 toddlers) or the regular therapy group (25 toddlers). The age group of infants/preschool children is selected based on the previous studies on early power mobility training in infants and preschool children. Power mobility training is typically offered to children between two and six years of age, with three years being the average age of the youngest child being recommended for a powered chair. However, studies showed that early power mobility training was feasible for 7-month-old infants and 18-month-old children with mobility disabilities. The participant's performance is indicative of the extent to which early power mobility training is feasible for both young infants and up to 3-year-old child with disabilities.

Recruitment: The children were recruited from self-referrals, health care practitioners, or the hospitals in Taipei and Taoyuan, Taiwan where children with motor delays (>1.5 sd) were receiving outpatient rehabilitation. The research team initially posted flyers describing the study at clinical settings and contacted the therapists in the clinical settings to introduce the goals,criteria and general procedure of the study. Parents/guardians obtained information about the study through the flyers and their therapists. Parents/guardians, who were interested and whose children met the criteria of diagnosis, age, capability determined by the doctor and their therapists, were given contact information for the investigator. After receiving contact information, the research team contacted the parents/guardian and/or therapists for scheduling a date of further testing by the research team at the hospital. When the research team contacted the parents, study was explained and parents received a letter detailing the procedure and given an opportunity to ask questions. Parents/guardians signed this informed consent form at the time of the first visit.

Procedure: Before the preintervention assessments, the research team will modify the car's seat and acceleration to the hand switch-driven, which allows the car to be derivable for the child who meets the inclusion criteria. Each child will have a customized ride-on toy car in the ROCBT and early powered mobility training groups. After modifications, they will receive preintervention assessments, including behavioral videotaping and developmental assessments. The developmental assessments will occur at the first and last week of the 9-week intervention, and the end of the 9-week follow-up phase. A therapist who does not involve in the intervention and is blinded to the study purpose will complete all the developmental tests. The driving and socialization behaviors will be videotaped by the research team for 1 hour/per session, one session/per week before, during and after the intervention phase at the hospital. In addition, participants will wear two accelerators on their wrists to monitor the physical activity during the 1 hour videotaping session. All videotapes will be coded by two independent coders, who are undergraduate students. Prior to making their ratings, the coder is instructed as to coding procedures by the PI, but he/she is not informed about the group assignment and the purpose of the study. Cohen's kappa coefficient will be calculated between the two independent raters to establish good reliability before formal coding.

Intervention: The research team will ask caregivers to identify goals (before intervention), and measure progress using goal-attainment scaling (GAS) before and after the intervention for the three groups. Ride-On Cars with Bi-manual Training Program (ROCBT): The research team will ask caregivers to identify goals (before intervention), and measure progress using goal-attainment scaling (GAS). Investigators will discuss with the clinical therapists who will provide training program in a hospital for 2 hours/per session, 2 sessions/per week for a total of 9-week intervention. Each week the research team will videotape the child's natural play and driving performance for the first hour of training session during the intervention phase. The 2-hour training session is composed of two 30-minute driving sessions and two 30-minute bi-manual training sessions. Each 30-minute driving training is followed by one 30-minute bi-manual training. Every week's treatment program will pre-planned and adjusted by the occupational therapist and the caregivers through discussion and clinical observation of participant's performance in the previous session. Training will still concentrate on building the concept of casual-effect on the switch and car motion, goal-oriented driving in a hospital, and bi-manual use in functional tasks for exploration in bi-manual training, discussed by the family, the treating therapist and the research team.

The car driving training includes 2 phases: I-car exploration and II-prompted driving. Participants can learn how to move and stop the car in the car exploration phase. Through prompted driving in phase II, they can use the car as a mean to explore environments (e.g., to the elevator, to different stores) and contact with people (e.g., drive to the caregiver and get the toy). Bi-manual training involves activities which include perceptual motor tasks (e.g., smear both hands with color), holding and manipulative tasks (e.g., cutting toy vegetables or fruits), posture and balance (e.g., pull a cart), and self-care and activities of daily living (e.g., drinking water from a cup with two handles).

Early Mobility Training Program: Most of the guidelines are similar with ROCBT, except for the bi-manual training. The therapist and family will merely focus on independent mobility training and improving socialization. The training time and period is the same as ROCBT.

Regular Therapy Program: The regular therapy group will continue the regular therapy, including physical, occupational and speech therapy. The general propose of the training is to improve the developmental scales, mobility, socialization and upper limb use in functional tasks. The research team will videotape the child's natural play and driving performance at the hospital for 1 hour/per session, 1 session/per week during the 9-week intervention phase.

Follow-up: This period will focus on the 9-week follow-up after receiving a treatment program. No treatment programs will be delivered to the participants. The research team will still videotape the child's natural play and driving performance at the hospital for 1 hour /per session, 1 session/per week during the 9-week follow-up phase.

Instrument and Procedure: Each participant will receive pre-intervention assessments, including behavioral videotaping and developmental assessments. Behavioral coding involved the mobility/driving performance during the 10-minute Car Play and socialization during the whole 20-minute Play (i.e., 10-minute Natural Play and 10-minute Car Play). The developmental assessments occurred at the first and last week of 9-week intervention, and the end of the 9-week follow-up phase, including the Pediatric Evaluation of Disability Inventory (PEDI), the Bayley Scales of Development, Peabody Developmental Motor Scales 2nd , Goal Attainment Scale (GAS), The Affordances in the Home Environment for Motor Development (AHEMD), and Parenting Stress Index (PSI). Necessary materials include two video cameras, a parent log and a customized ride-on car.

Data Reduction and Analysis: All videotapes will be coded by two independent coders, who are undergraduate students. Prior to making their ratings, the coder is instructed as to coding procedures, but he/she is not informed about the group assignment and the purpose of the study.

Mobility Measures: The following measures will be obtained via video coding the 10-minute Car Play during pre-intervention, intervention and post-intervention phases to determine the feasibility of learning to drive the car:

1. Driving Categories (time in seconds): a. Independent Mobility: When the child independently drives the car preceded by an independent switch contact without an adult's assistance. b. Assisted Mobility: When an adult puts the child's hand on the switch but he independently pushes the switch to begin driving. c. Caregiver Mobility: When the child drove with an adult's hand directly on top of his hand.
2. Visual Attention to Switch: The frequency (number of times) that the child looked at the switch during the 10-minute driving.
3. Stopping Categories (number of times divided by total times goal was presented): a. Independent Stop: When the child independently moves his hand off the switch and makes the car stop within one car length of the goal location. b. Stops with Verbal Cues: When the child moves his hand off the switch as the car arrives the goal only after verbal cues given from an adult. c. Stops with Tactile Contacts: When the child moves his hand off the switch as the car arrives the goal only after tactile cues (e.g., touching his hand or moving his hand off the switch) given from an adult.

Socialization Measures: To examine the impact of independent mobility on the socialization during the 10- minute Natural Play and 10-minute Car Play, the following measures will be obtained via coding video footage during pre-intervention, intervention and post-intervention:

1. Reaching for toy/person: The frequency (number of times) that the child initially extends arms to the play toy/interacting person.
2. Initiation of contact with others: peer-directed or adult-directed: Target child-initiated contacts with others are counted whenever two conditions are met: (a) the target child initiates the contact with another individual without any observable prompting or initiating behavior on the part of another person and (b) the target child independently vocalizes (with either comprehensible words or other vocalizations, including shouting, laughing, grunting, etc.) or physically points to, touches, or indicates that he or she wants something from another individual. Target child-initiated contacts and vocalizations are divided into two categories: (i) peer-directed and (ii) adult-directed.
3. Other initiated contacts: contact by peers or by adults: Peer-initiated contacts are defined as any child initiating any type of contact with the target child (e.g., talking to the child, touching the child or a mobility device the child is using, giving a toy or item to the child, taking a toy or item away from the child). Adult-initiated contacts with the target child are: (a) carrying, moving, or otherwise touching the child or the device in which the child is seated (e.g., swing, wheelchair, toy car); (b) taking a toy or item away from the child.
4. Facial Expression: The frequency (number of times) of both positive and negative facial expressions appeared during interaction. Positive was determined to include smiling and laughing. Negative was determined to include discomfort, crying and unhappy facial expression.
5. Vocalization/Gesture: The frequency (number of times) that the child vocalizes/gestures to a play toy or person, including grunting, shouting, vowel-type sounds (e.g., ee, i, ah, oo u).

Repeated measure one way ANOVA will be used to compare the mean difference of using a toy car for mobility, socialization and development before and after the intervention, and after 9-week follow-up, i.e., within group comparison. One way ANOVA will be used to compare the mean difference of all developmental tests (mobility, socialization, motor, and cognition), participation and physical activity for exploration among three groups before and after the intervention and the end of follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

1. motor delays (sd>1.5) resulting in motor impairments that prevented functional independent mobility, such as rolling, crawling, walking;
2. aged between 12 months to 36 months old
3. able to tolerate sitting with support for 30 minutes
4. able to reach the objects with either one or two hands
5. consent of the parents to agree to the testing procedures and participate in the training program at the hospital.

Exclusion Criteria:

1. children with severe sensory impairments such as blindness, deafness
2. parents/caregivers are not able to make a time commitment for the training phase

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in General Mobility and Social Development at 9 weeks and 18 weeks as assessed by the Pediatric Evaluation of Disability Inventory (PEDI) | Assessment will occur 3 times during the whole study, including the first and last week of the 9-week intervention, and the end of the 9-week follow-up phase.
  PEDI is a set of tests for children from 8 months to 6 years old. The PEDI quantified self-care, mobility, and social functions. The PEDI is especially useful for tracking changes in functional skills.
Mobility/Driving Performance as assessed by the coding behaviors from the videotaping | The driving behaviors will be followed for the duration of implementing the intervention program at the hospital, an expected average of 9 weeks.
  The driving behaviors will be coded from each 10-minute Car Play session: a) amount of time moving/total time, b) frequency, time and duration of parental assistance (physical and/or vocal), c) number of successful "directional driving trials". In each of 10 trials, the child is asked to drive 5 feet to the parent or researcher. He/she is given 30 seconds to complete the distance and make a stop at the goal.
Socialization as assessed by the coding behaviors from the videotaping | The socialization behaviors will be followed for the duration of implementing the intervention program at the hospital, an expected average of 9 weeks.
  The frequency and duration related to socialization will be coded during the whole 20-minute Play, including 10-minute Natural Play and 10-minute Car Play: physical contacts, initiation of contact with others, other initiated contacts, facial expressions, vocalizations/gestures and mutual play events (ex. sharing a toy).
Physical activity as assessed by the amount of counts from the wrist accelerometers | The physical activity will be recorded for the duration of implementing the intervention program at the hospital, an expected average of 9 weeks.
  Each week the participant will wear the accelerometers on both wrists during the 1 hour videotaping session, including 30-minute driving and 30-minute natural play. The accelerometers code the physical activity for driving and playing.

SECONDARY OUTCOMES:
Change from baseline in General Development at 9 weeks and 18 weeks as assessed by The Bayley Scales of Development | It will be administered a total of 3 times during the whole study, including the beginning and end of the 9-week intervention, and the end of the 9-week follow up.
  GAS is family-centered, criterion-referenced and responsive tool. There are 5 possible outcomes: a score of 0 means the child has attained the goal, whereas scores of -2 and -1 represent lower than expected performance and +1 and +2 are higher than expected performance.
Change from baseline in General Development at 9 weeks and 18 weeks as assessed by the Goal Attainment Scale (GAS) | It will be administered a total of 3 times during the whole study, including the beginning and end of the 9-week intervention, and the end of the 9-week follow up.
  GAS is a family-centered, criterion-referenced, reliable, valid and responsive tool. There are 5 possible outcomes: a score of 0 means the child has attained the goal, whereas scores of -2 and -1 represent lower than expected performance and +1 and +2 are higher than expected performance.
Change from baseline in General Development at 9 weeks and 18 weeks as assessed by the Affordances in the Home Environment for Motor Development (AHEMD) | It will be administered a total of 3 times during the whole study, including the beginning and end of the 9-week intervention, and the end of the 9-week follow up.
  AHEMD is a reliable and valid assessment to assess the quality and quantity of motor development opportunities in the home during early childhood. Age-related AHEMD questionnaires were developed (3-to-18 months; and 18-to-42 months) and translated into four different languages: English, Chinese Portuguese, and Spanish. Test-retest reliabilities for AHEMD-Toddler-C were adequate (0.46~0.93). For convergent validity, the correlation coefficients between AHEMD and Home Observation for Measurement of the Environment Inventory (HOME) were 0.44.
Change from baseline in Parents' Perceptions at 9 weeks and 18 weeks as assessed by Parenting Stress Index (PSI) | It will be administered a total of 3 times during the whole study, including the beginning and end of the 9-week intervention, and the end of the 9-week follow up.
  PSI is a tool that was designed to measure the overall level of parenting stress experienced by parents of children between the ages of one month and twelve years.
The Revised Dimensions of Mastery Questionnaire (DMQ 18) - Chinese version | it will be administered a total of 3 times during the whole study, including the beginning and end of the 9-week intervention, and the end of the 9-week follow up.
  The Revised Dimensions of Mastery Questionnaire (DMQ 18) - Chinese version: was used to measure both instrumental and expressive aspects of mastery motivation by caregiver report. There are 7 scales (cognitive/object persistence, gross motor persistence, social mastery motivation with adults, social mastery motivation with children/peers, mastery pleasure, negative reactions to challenge in mastery situations, and general competence) and Likert-type items rated 1-5(from not at all like this child to exactly like this child). The DMQ 18 contained four parallel age-related versions for children aged 6 months to 19 years (infant, preschool, school-age rated by adults, and school-age self-report). The DMQ 18 show good internal consistency (.72-.96). The intra- and inter-rater reliability were acceptable for the DMQ18 (ICCs=0.61-0.87).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Huang HH, Chen YM, Huang HW, Shih MK, Hsieh YH, Chen CL. Modified Ride-On Cars and Young Children with Disabilities: Effects of Combining Mobility and Social Training. Front Pediatr. 2018 Jan 15;5:299. doi: 10.3389/fped.2017.00299. eCollection 2017. PMID 29387682